CLINICAL TRIAL: NCT05736692
Title: Addressing Sleep in Adolescents Post-Concussion ("ASAP Study"): A Phase 2 Clinical Trial
Brief Title: Addressing Sleep in Adolescents Post-Concussion ("ASAP Study")
Acronym: ASAP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Despite intensive recruitment efforts, we have been unsuccessful enrolling participants. Study being halted due to futility.
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-0608
Record Dates: First submitted 2023-02-11; First posted 2023-02-21 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Concussion, Brain; Sleep Disorder
MeSH Terms: conditions — Brain Concussion; Sleep Wake Disorders

STUDY DESIGN:
Intervention Model Description: This is a straightforward two-arm parallel randomized clinical trial with follow-up 1 week and 1 month post-randomization. Eligible adolescents will participate for up to 5 weeks. Week 1 will involve pre-randomization sleep monitoring, and will conclude with a study visit during which staff will review sleep data and give measures of PPCS severity and other outcomes. At that visit, youth who have both PPCS and poor sleep quantity or quality will be evenly randomized to receive the intervention or continue care-as-usual (control). Short-term and extended follow-up assessment will occur in Weeks 2 and 5.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Sleep Intervention (Experimental): 1-session intervention designed to improve adolescent sleep quality and/or quantity.
  Interventions: Behavioral: Brief Sleep Intervention
- Control (No Intervention): Care as Usual. Those in this condition will be asked to continue their scheduled/prescribed care until the next study assessment. Note that, to ensure that all participants (control and sleep intervention) are offered the current standard of care, all will get a simple handout on sleep hygiene and any who is not receiving follow-up care will be referred to the Brain Health and Wellness Center (the multidisciplinary program to which all PCSS care at Cincinnati Children's is routed).

INTERVENTIONS:
Behavioral: Brief Sleep Intervention — A ~50-minute semi-structured intervention based on the behavioral sleep medicine literature, particularly for adolescent insomnia, focused on key elements that can be addressed in one session. Treatment elements include engaging motivation, goal setting, barrier identification, problem-solving, pre-planning, self-monitoring, and setting rewards. The interventionist will be sensitized to barriers to sleep quality and quantity particularly relevant during adolescence, including job/work, homework, and social obligations, use of nicotine and caffeine, and social media and electronic devices. The interventionist will converse primarily with the adolescent, but parents will remain in the room as a support in problem-solving and executing therapeutic plans.
  Arms: Brief Sleep Intervention

SUMMARY:
Hundreds of thousands of adolescents experience protracted recoveries from concussion, which can affect all aspects of their lives and create family and societal burden. Research suggests that interventions to improve their sleep quantity and/or quality could improve recovery from concussion, but current treatment models are costly and onerous for families, fit poorly with integrated care models, and leave youth and their families to suffer months of protracted burden. This study will evaluate the efficacy of a promising brief behavioral sleep intervention, which could prove to be a powerful new tool to head off protracted symptom burden.

DETAILED DESCRIPTION:
Over 500,000 adolescents sustain mild traumatic brain injuries (aka "concussions") in the US each year. Despite the term "mild," concussion symptoms disrupt all aspects of an adolescent's functioning, from school to friendships to family, and impair quality of life. Although many youth recover quickly, ~1/3 still have protracted postconcussive symptoms (PPCS) a month or later post-injury. PPCS are hard to treat medically, as concussion-induced pathophysiology wanes within 1-3 weeks. Instead, contemporary treatments seek to target modifiable patient behaviors that contribute to PPCS. There is accumulating evidence that poor sleep quality or quantity are under-addressed, potent, treatable contributors to PPCS, particularly for adolescents. Indeed, recent studies suggest that targeted behavioral sleep treatments can improve adolescent sleep and other persistent post-concussive symptoms, but published approaches have required 4-6 treatment sessions delivered months post-injury. Such approaches are costly and onerous for families, fit poorly with integrated care models, and leave youth and their families to suffer months of protracted PPCS burden. In contrast, our team has developed a single-session behavioral sleep intervention for adolescents that is designed to be delivered soon after acute pathophysiology wanes (4-7 weeks post-injury) to head off protracted symptom burden. Preclinical and Phase 1 studies suggest that this approach is feasible, well-accepted, and has the potential to improve both sleep and other PPCS. Our long-term plan is to test the effectiveness of that intervention in an applied setting. To justify and guide that large-scale trial, here we propose a Phase 2 clinical trial to definitively test the efficacy of the intervention in a controlled context. We will randomize 70 adolescents aged 12-18 years who are experiencing PPCS and poor sleep quantity or quality to receive either a 1-session sleep treatment (Tx) or care-as-usual (control) 4-7 weeks post-injury. We will assess sleep, PPCS, and real-world functioning just prior to randomization and then again 1 week and 1 month later. Our primary aim is to determine the short-term efficacy of the Tx in improving both sleep and PPCS. Secondarily, we will assess the sustained efficacy of the Tx and its impact on daily functioning. We will also explore potential effect modifiers (e.g., demographics, injury-related factors). To ensure successful completion of this study, we have assembled a team of experts in pediatric brain injury and PPCS, adolescent sleep research, behavioral sleep medicine, and biostatistics with a proven record of successful collaboration, including on similar studies and our Phase 1 trial. The current study represents an important next step in our research program, definitively testing efficacy in a Phase 2 trial prior to embarking on a larger (Phase 3) applied effectiveness study. If, as we propose, our brief intervention both improves sleep and reduces other PPCS, this could lead to a powerful new tool to accelerate the recovery and alleviate burden for hundreds of thousands of adolescents every year.

ELIGIBILITY:
Inclusion Criteria:

Had a concussion resulting in at least one persisting symptom at study entry 3-6 weeks later (initial visit 4-7 weeks post-injury). Those with Persistent Post-Concussive Symptoms (PPCS) and poor sleep at the initial visit will be eligible for randomization. PPCS will be defined as: concussion (blow to the head with loss of consciousness <30 min, amnesia, or alteration in mental status) resulting in >1 new symptom on the Post-Concussion Symptom Scale that persists at at least 4 weeks post-injury. Poor sleep quantity or quality will be defined as: (a) objective actigraphy showing less than recommended sleep (<8 hours) on school nights or spending <85% of the sleep period actually asleep, or (b) self-report of poor sleep quality (score >5 on the Pittsburgh Sleep Quality Index).

Exclusion Criteria:

(a) lowest injury-related Glasgow coma scale (GCS) <13 or imaging evidence of intracranial abnormality, (b) previous more severe TBI or previous mTBI from which recovery was incomplete, (c) associated extracranial injury that could persistently impact sleep (e.g., due to immobility), (c) non-fluent in English, (d) previously-diagnosed intellectual disability, autism, bipolar disorder, or psychosis, (e) not attending in-person or virtual school requiring morning attendance, (f) use of medication known to substantially affect sleep (e.g., stimulant).

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Objective Sleep Assessment | Measured during the week leading up to each of the three study visits
  Youth will wear a wrist-based actigraph/accelerometer and report sleep-wake patterns on a nightly sleep diary. This low-burden approach tracks sleep in the natural setting and yields objective estimates that have >90% agreement with EEG-defined sleep in adolescents. Following the PI's established protocols, during the assessment portion of each visit, study staff will review the uploaded data and sleep diary conjointly with the parent and youth to identify and exclude artifacts (e.g., unit removal). The primary sleep endpoints (Aims 1-3) will be sleep period on weeknights (onset to offset) and percent of that period actually spent asleep.
Persistent Post-Concussive Symptom Severity | Measured at all three study visits
  The Post-Concussion Symptom Scale (PCSS) is a well-validated self-report form that asks about the presence/severity of 22 symptoms. Consistent with prior recovery studies, youth will be asked to endorse only those items that started at the time of injury and persist. The primary PCSS severity endpoint (Aims 1-3) will be total score, excluding items asking about sleep.
Overall Daily Functioning | Measured at all three study visits
  Parent- and self-report on the 23-item Pediatric Quality of Life (PedsQL generic) questionnaires. The PedsQL has extensive psychometric support in children and adolescents with a variety of conditions, is a suggested common data element in TBI research, and is sensitive to adolescent PPCS. The primary daily functioning endpoints (Aims 2 & 3) will be parent- and self-report PedsQL total scores.

CONTACTS AND LOCATIONS:
Overall Officials: Dean W Beebe, Ph.D., Principal Investigator — Cincinnati Children's
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon publication of primary analyses (or within 2 years of study completion in the unlikely event of no such publication), we will have available the Final Dataset that has been de-identified in a HIPAA-compliant fashion and carefully reviewed to make sure that non-HIPAA-designated but potentially identifying information are not included (e.g., rather than have dates of birth and participation, we will include the more analytically-relevant variable of exact age). Descriptors for all variables shared will be included to prevent misuse or confusion. The Final Dataset will be provided at no charge to qualified individuals requesting it from the PI. We also plan to provide relevant aspects of the dataset as a secondary file attached to the online version of the primary publication.
Supporting Information: Study Protocol, ICF
Time Frame: Upon publication of primary analyses (or within 2 years of study completion in the unlikely event of no such publication), data will become available. We expect that such access will extend at least 5 years beyond completion of the study.
Access Criteria: Final Dataset will be provided at no charge to qualified individuals requesting it from the PI.